CLINICAL TRIAL: NCT03936231
Title: ASSESSMENT OF THE MECHANICAL POWER TRANSMITTED TO THE PATIENTS WITH MECHANICAL VENTILATION IN INTENSIVE CARE UNITS "MECHANICAL POWER DAY"
Brief Title: Cross-sectional, Observational, Prospective and Analytical Study:MECHANICAL POWER DAY (MPDay)
Acronym: MPDay
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hospital Universitario Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Alejandro Gonzalez Castro, Critical Care Department, Hospital Universitario Marqués de Valdecilla
Other Study IDs: 2019.040
Record Dates: First submitted 2019-04-24; First posted 2019-05-03 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Mechanical Ventilation Complication
Keywords: VILI; Mechanical Power; Driving Pressure; Strain; Stress
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NO Intervention — Given the observational nature of this study, we consider that no intervention is required.
  Participation in concomitant studies: given the observational condition of this study, patiens that are included in other observational and/or experimental researches, can be included in the current study.

SUMMARY:
Recently the new concept of "mechanical power" has been proposed. It refers to the amount of energy per minute that is transferred to the lung by the ventilator. The generation of this form of energy would include both parameters that were previously proposed to be possible causes for lung damage and new parameters that had not been taken into account until now, such as the flow rate or the respiratory rate, without forgetting the individual characteristics of each ventilated subject.

The main objective of the current study is to know the value of the mechanical power in the patient connected to mechanical ventilation, in a volume control model.

This value will be calculated from electronically provided data using the simplified formula by Gattinonni et. al.

DETAILED DESCRIPTION:
Introduction and justification:

Over the last few years the investigators have witnessed an important technological developement in the field of mechanical ventilation. Along with the technological advances, the better understanding of the respiratory physiopathology has shown that mechanical ventilation "per se" can lead to deleterious effects.

In this context, the search for those variables which are responsible for the developing of ventilator-induced lung injury (VILI) has become an important goal in this field. In fact, the investigators are witnessing the nearly exponential increase in the publication of studies that have tried to associate the different parameters that intervene in mechanical ventilation with the injury to the lung structure.

Recently the new concept of "mechanical power" has been proposed. It refers to the amount of energy per minute that is transferred to the lung by the ventilator. The generation of this form of energy would include both parameters that were previously proposed to be possible causes for lung damage and new parameters that had not been taken into account until now, such as the flow rate or the respiratory rate, without forgetting the individual characteristics of each ventilated subject.

12J/min has been stablished experimentally as the energy threshold from where changes in the lung that can lead to VILI begin to appear. Nevertheless, the true issue would be to get to know the best way to normalize the mechanical power value. However, it seems reasonable to think that the values of energy originating VILI in experimental animal models and in humans are different.

Nowadays, in spite of the wide range of monitoring systems that the investigators have, the investigators still don´t know the real mechanical power that the investigators are transmitting to our patients. The different research teams that have deepened into the subject have seen themselves forced to infer their results from retrospective data and from very selected samples of patients immersed in different studies. As one of the first steps in the way of a better understanding of the impact of "mechanical power", the investigators believe it is justified to develope a descriptive and observational study to get to know the real mechanical power value the investigators ventilate our patients in the ICU with.

Objective and hypothesis:

Clinical guides and recommendations aimed at improving ventilation basing on the characteristics of the different pathologies in order to minimize VILI do exist, but the fact remains that the threshold of mechanical power in mechanical ventilation is still unkown.

The main hypothesis of the present study is that the mechanical power received by the patients who need mechanical ventilation in the intensive care unis is greater tan the threshold that has been established by experimental models.

Moreover, the investigators think that mechanical power varies considerably depending on the current and previous pathology of the patient and the days on mechanical ventilation.

Resting on the previous hypothesis, the main objective of the current study is:

- Know the value of the mechanical power in the patient connected to mechanical ventilation, in a volume control model.

This value will be calculated from electronically provided data using the simplified formula by Gattinonni et. Al.

Secondary objectives are:

* Analyze the epidemiology of different modalities in ventilatory, not just VC, on the basis of the collected variables.
* To assess if the transmitted mechanical power varies depending on the pathology, on the days on mechanical ventilation or on the reason that leads to the need for mechanical ventilation.
* In case of a ventilatory mode which allows spontaneus breathing, the investigators can see the variability of the plateau pressure and if the investigators can infer its value in the calculation of mechanical power.
* To know the driving pressure and the ventilatory ratio of ventiled patients.
* To establish differences among the main analysed parameters depending on the type of critical carea area studied.

Design and methodology:

Cross-sectional, observational, prospective and analytical study. The variables of the study will be collected on a fixed date as agreed with the participating ICU. These variables will be registered during the period of time between 8 am to 15 pm on the 21st of November 2019, in order to adjust to the normal working routine at an intensive care unit.

Sample selection:

All patients that are hospitalised in a critical care unit and on mechanical ventilation on the 21st of November 2019.

Inclusion criteria:

All the patients hospitalised in a crital care unit who are on invasive mechanical ventilation, whatever the cause.

ELIGIBILITY:
Inclusion Criteria:

* Patiens with mechanical ventilation in the critical care areas.

Exclusion Criteria:

* Patients with not mechanical ventilation.
* Patients with mechanical ventilation for less that 6 hours.
* Traqueostomy patients
* APRV or BiLEVEL ventilation mode.
* Noninvasive ventilation d.n selectiv
* Selective ling ventilation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that are hospitalised in a critical care area and on mechanical ventilation on the 21st of November 2019.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2019-11-21 (Estimated); Primary Completion 2019-11-21 (Estimated); Study Completion 2019-11-21 (Estimated)

PRIMARY OUTCOMES:
Mechanical Power (MP) (assess the amount of energy per minute that is transferred to the lung by the ventilator) | One Day
  MP=0.098 x Vt x Fr x Pp-(Pplat-PEEP/2)

CONTACTS AND LOCATIONS:
Locations (1):
- Alejandro Gonzalez-Castro, Santander, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Castro A, Medina Villanueva A, Escudero-Acha P, Fajardo Campoverdi A, Gordo Vidal F, Martin-Loeches I, Rocha AR, Romero MC, Hernandez Lopez M, Ferrando C, Protti A, Modesto I Alapont V; Mechanical Power Day Group. Comprehensive study of mechanical power in controlled mechanical ventilation: Prevalence of elevated mechanical power and component analysis. Med Intensiva (Engl Ed). 2024 Mar;48(3):155-164. doi: 10.1016/j.medine.2023.11.004. Epub 2023 Nov 22. PMID 37996266